CLINICAL TRIAL: NCT06319950
Title: High-dose Furmonertinib Versus Osimertinib as First-line Treatment in Advanced EGFR Mutation-positive NSCLC Patients With Brain Metastases: a Multi-center, Randomized, Controlled, Prospective, Phase II Clinical Trial
Brief Title: High-dose Furmonertinib Versus Osimertinib in Advanced EGFRm NSCLC Patients With Brain Metastases
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Dongqing Lyu, MD, Chief Physician, Taizhou Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20240229
Record Dates: First submitted 2024-03-01; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer, Nonsmall Cell
Keywords: non-small cell lung cancer (NSCLC); brain metastases; epidermal growth factor receptor (EGFR); tyrosine kinase inhibitors (TKI)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — aflutinib; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-dose Furmonertinib group (Experimental): Furmonertinib, 160mg po qd
  Interventions: Drug: Furmonertinib
- Osimertinib group (Active Comparator): Osimertinib, 80mg po qd
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Furmonertinib — Furmonertinib, 160mg po qd
  Other Names: AST2818; alflutinib
  Arms: High-dose Furmonertinib group
Drug: Osimertinib — Osimertinib，80mg po qd
  Other Names: AZ9291
  Arms: Osimertinib group

SUMMARY:
The investigators were to explore whether high-dose Furmonertinib, compared with osimertinib, could achieve longer survival in patients with EGFR-mutated NSCLC with CNS metastasis.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer incidence and death worldwide. Non-small cell lung cancer accounts for about 80-85%, and EGFR mutations occur in about 45-55% of the Asian population. In newly diagnosed NSCLC patients, the rate of brain metastases in advanced NSCLC can be as high as 25% to 44%. The brain metastasis rate of advanced lung adenocarcinoma with EGFR mutation can reach 60%. For NSCLC patients with CNS metastases and EGFR mutations, the PFS of EGFR-TKIs was improved compared with chemotherapy, but neither was satisfactory, even with Osimertinib (third-generation EGFR-TKI). The PFS of patients with CNS metastases treated with Osimertinib was only 15.23 months. Therefore, the diagnosis and treatment of lung cancer patients with brain metastases is still a difficult problem to improve the long-term survival rate of lung cancer. Clinical data and early preclinical studies have shown that Furmonertinib(AST2818) can effectively inhibit the classical mutation of EGFR, especially for intracranial lesions, and is well tolerated. In the FURLONG study, the PFS of patients with CNS metastases was 20.8 months and the ORR were 91%, respectively. This may be due to the unique molecular structure of Furmonertinib, which has the advantage of "double entry into the brain". Furthermore, the investigators' previous research showed that patients treated with 160mg of Furmonertinib after third-generation EGFR-TKIs treatment resistance were divided into intracranial progression mode group and extracranial progression mode group, and finally proven that Furmonertinib 160mg with or without antiangiogenic agents could be an option for patients with advanced NSCLC who have developed resistance after third-generation EGFR-TKIs, especially those who have developed resistance due to intracranial lesion progression. Based on above, the investigators propose to develop a multi-center, randomized, controlled, prospective, Phase II clinical trial in order to explore whether high-dose Furmonertinib could achieve longer survival in patients with EGFR-mutated NSCLC with CNS metastasis, particularly long-term control of intracranial lesions.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged >=18 and <=80 years old.
* Patients with histologically or cytologically confirmed NSCLC with adenocarcinoma or adenocarcinoma components predominant, and with central nervous system metastases (with measurable lesions).
* The tissue or blood sample is determined to be EGFR positive (including rare EGFR mutations) by testing by a tertiary Class A hospital or a qualified testing institution, and the tissue submitted for testing cannot be from a tumor lesion that has been treated with radiation, but can be used for a new lesion after local treatment.
* Patients who had not previously received systemic anti-tumor therapy for locally advanced or metastatic non-small cell lung cancer (patients who had received first-line chemotherapy but had not received TKIs could be enrolled). Patients who have undergone radical surgery, radical chemo-radiotherapy, or adjuvant therapy (chemotherapy, radiation) for early NSCLC may be enrolled if they later develop disease recurrence or metastasis.
* Stable brain metastases that do not require local treatment of brain metastases either immediately or planned during the study period.
* According to RECIST v1.1, enrolled patients should have at least one tumor lesion in all tumors that can meet the following requirements: they have not been treated with local therapy such as radiotherapy in the past, and can be accurately measured at baseline, and the longest diameter at baseline is ≥10mm (in the case of lymph nodes, the short diameter is ≥15mm). Lesions that have previously received local treatment (radiotherapy or other treatment) can only be measured if disease progression occurs more than 6 months after the end of treatment.
* ECOG PS 0-1, and with no deterioration during the first 2 weeks of the study and expected survival time of no less than 3 months.
* Patients should have sufficient bone marrow reserve function, and no liver, kidney, coagulation dysfunction, laboratory test values must meet the following conditions:

  1. Absolute neutrophil count ≥ 1.5×109/L, and white blood cell count ≥3×109/L;
  2. PLT ≥100×109/L;
  3. Hb ≥90g/L;
  4. Serum Cr ≤1.5×ULN and eGFR ≥50 mL/min;
  5. AST and ALT≤2.5×ULN (or AST and ALT≤5×ULN for patients with liver metastasis)
  6. In the absence of proven liver metastasis, TB ≤1.5×ULN (or TB ≤3×ULN for patients with liver metastasis or Gilbert syndrome;
  7. INR ≤1.5, and APTT ≤1.5×ULN.
* Male patients and female patients of reproductive age should take adequate contraceptive measures within 3 months after signing the study informed consent to the last study drug treatment; In women of childbearing age, pregnancy test results are negative within 7 days before the first dose.
* All previous treatment-related toxicities (except alopecia and grade 2 neurotoxicity associated with previous platinum chemotherapy) had been recovered (to ≤ grade 1) before first administration of the investigational drug.
* The subject is able to understand and voluntarily sign a written informed consent (which must be signed prior to performing any procedure specified in the study protocol).
* Be able to voluntarily complete the study procedures and follow-up examinations as required by the study protocol.

Exclusion Criteria:

* Patients with the following treatments:

  1. Previous use of any EGFR TKIs therapy;
  2. Previously received systemic antitumor therapy (such as targeted therapy, biotherapy, immunotherapy, etc.) for advanced/metastatic non-small cell lung cancer;
  3. Standard chemotherapy within 28 days before the first administration of the study drug; The study received anti-tumor therapy with traditional Chinese medicine within 7 days before the first administration of the drug;
  4. Previous WBRT; Had received >30% of bone marrow radiotherapy or extensive radiotherapy within 28 days prior to the first dose of the study drug; Local radiotherapy (e.g., thoracic and rib radiotherapy) or palliative radiotherapy for bone metastases within 7 days prior to initial administration of the study drug;
  5. Uncontrolled pleuroperitoneal effusion and pericardial effusion;
  6. Uncontrollable cancerous pain; Anesthetic painkillers did not reach a stable dose at the time of enrollment;
  7. Study major surgery within 28 days before the first administration of the drug ( major surgery refers to grade 3 and grade 4 surgery in Measures for the Clinical Application of Medical Technology in China, on May 1, 2009 );
  8. Has received a strong inducer or suppressor of CYP3A4 within 14 days prior to initial administration of the investigatory drug or requires continued treatment during the study period (including Chinese herbal medicine, see Appendix for a list of drugs);
  9. Patients who are receiving and require continued treatment during the study with drugs known to prolong the QTc interval or that may cause tip torsion ventricular tachycardia (see Appendix for a list of drugs);
  10. Participants who have participated in other clinical trials within 28 days prior to the first administration of the investigational drug (except non-interventional drug trials);
* Patients with primary malignant brain tumors and unstable brain metastases. Definition of unstable brain metastases: Patients with CNS complications who require emergency neurosurgical treatment (such as surgery); Patients with an equivalent dose of dexamethasone or more than 5mg of glucocorticoids, mannitol or diuretics to control symptoms of brain metastases should be administered within 14 days prior to the first dose; The first study looked at patients who had received local radiotherapy or gamma knife treatment within 14 days prior to administration. Patients with meningeal metastasis were excluded.
* Patients who have had or have a history of other malignancies within the past 5 years (except cured basal cell or squamous cell carcinoma of the skin, papillary carcinoma of the thyroid gland, carcinoma in situ of the cervix, and ductal carcinoma in situ of the breast).
* The patient had symptoms of spinal cord compression caused by the tumor.
* Clinically significant gastrointestinal dysfunction that may affect the intake, transport, or absorption of investigational drugs, such as inability to take oral drugs, difficult to control nausea or vomiting, a history of extensive gastrointestinal resection, Untreated recurrent diarrhea, atrophic gastritis (onset age less than 60 years), untreated stomach disease requiring long-term use of PPI acid suppressants, Crohn's disease, ulcerative colitis.
* Cardiovascular and cerebrovascular diseases/symptoms/indications that meet any of the following conditions:

  1. Average resting QTc≥470ms (corrected QT interval, calculated according to Fridericia's formula, see Appendix 18-9), the average QTc of 3 ECG intervals of more than 5 minutes, and the QT interval should be measured from the beginning of the QRS complex wave to the end of the T wave;
  2. Any abnormalities in rhythm, conduction, or morphology of the clinically significant resting ECG, such as complete left bundle branch block, 2nd and 3rd degree heart block, PR interval > 250ms;
  3. Any factors that increase the risk of prolonged QTc or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or sudden unexplained death in a first-degree relative under the age of 40-year-old, or any combination of medications known to prolong the QT interval;
  4. LVEF <50%;
  5. Patients with a history of decreased myocardial contractility and related symptoms in the 6 months prior to study administration, such as chronic congestive heart failure, pulmonary edema, or decreased ejection fraction;
  6. Patients with a history of acute and chronic cardiovascular and cerebrovascular disease and related symptoms within 6 months prior to study administration, such as myocardial infarction, severe or unstable angina pectoris, cerebral infarction, cerebral hemorrhage, or transient ischemic attack.
* Persons infected with HIV, syphilis, HCV or HBV, meeting the following conditions:

  1. HBs Ag positive and HBV DNA ≥2000cps/ mL (or 500IU/ mL);
  2. Anti-HCV antibody and HCV RNA positive;
  3. HIV antibody positive.
* Prior or screening history of interstitial lung disease or ILD, or drug-induced ILD, or radiation pneumonia requiring hormone therapy, or any evidence of active ILD (such as acute onset or progressive pneumonia/pulmonary fibrosis at baseline), or pulmonary symptoms deemed unsuitable for inclusion by the investigator or risk factors deemed unsuitable for interstitial lung disease.
* Had previously received allogeneic bone marrow transplantation.
* Pregnant and lactating women.
* The patient has any other disease or medical condition that is unstable or may affect their safety or study compliance, any serious or uncontrolled systemic disease, including autoimmune disease requiring corticosteroid therapy, uncontrolled hypertension (SBP ≥150 mmHg or DBP ≥95 mmHg), Uncontrolled diabetes, active bleeding, eye lesions, and other serious mental, neurological, cardiovascular, or respiratory diseases.
* Known or suspected allergy to the investigational drug ingredient or its analogues.
* The subjects were judged by the investigator to be unfit for this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival(PFS) | 5 years from first patient randomized.
  The time from the start of randomization until the first occurrence of disease. progression or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
objective response rate(ORR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The proportion of patients with a complete or partial response
Intracranial objective Response Rate(iORR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The proportion of patients with a complete or partial response of intracranial tumors
Intracranial progression free survival(iPFS) | 5 years from first patient randomized.
  The time from the beginning of randomization to the first occurrence of objective progression or death of intracranial tumors, whichever occurs first.
overal survival time(OS) | 5 years from first patient randomized.
  The time from randomization to death from any cause
Disease control rate(DCR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  the proportion of patients with a complete response, partial response, or stable disease
Intracranial disease control rate(iDCR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  the proportion of patients with a complete response, partial response, or stable disease(≥6w) of intracranial tumors
Depth of response (DepOR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  best percentage change in the sum of the longest diameter of target lesions compared with baseline in patients without progression of non-target lesions and the occurrence of new lesions
Depth of intracranial response(iDepOR) | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  best percentage change in the sum of the longest diameter of target lesions in CNS compared with baseline in patients without progression of non-target lesions and the occurrence of new lesions
Time to intracranial remission(iTTR) | 5 years from first patient randomized.
  The time from randomization to the first assessment of CR or PR for intracranial tumor.
Duration of response(DoR) | 5 years from first patient randomized.
  The time from the date of first documented response to the date of disease progression or death, whichever occurred first.
Duration of intracranial response(iDoR) | 5 years from first patient randomized.
  The time from the date of first documented response in CNS to the date of disease progression or death, whichever occurred first.
Rate of improvement in neural function | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  Changes in Karnofsky scores and neuro-oncology Scale scores from baseline
Health-related quality of life | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  Changes in FACT-L scale scores from baseline
Adverse events | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The type, frequency, severity, and degree of treatment-related adverse events (according to CTCAE version 5.0)

OTHER OUTCOMES:
Dynamic changes of ct-DNA | Duration of time from the start of treatment to the end of study, assessed up to 5 years
  The dynamic changes of ct-DNA in patients' blood before and after 3 weeks of medication